CLINICAL TRIAL: NCT03731936
Title: Artificial Intelligence to Assess the Association Between Facial Characteristics and Coronary Artery Diseases
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 20181104-2017-907
Record Dates: First submitted 2018-11-04; First posted 2018-11-06 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease
Keywords: artificial intelligence; facial characteristics
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Model establishment and test group: Patients undergoing coronary angiography or coronary computer tomography angiography will be enrolled. Patients data will be used to establish the facial based diagnostic model of coronary artery diseases, and to prospectively validate the diagnostic effectiveness of the model.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purposes of this study are 1) to explore the association between facial characteristics and the increased risk of coronary artery diseases; 2) to evaluate the diagnostic efficacy of appearance factors for coronary artery diseases.

DETAILED DESCRIPTION:
Several age-related appearance factors were described associated with increased risk of coronary artery diseases (CAD). However, several limitations made these facial risk factors hard to be utilized in clinical practice, including 1) low prevalence in CAD patients, 2) lack of specific definition, 3) poor reproducibility in artificial recognition.

Thus, the investigators designed a multi-center, cross-sectional study to explore the association between facial characteristics and CAD and evaluate the diagnostic efficacy of appearance factors for CAD. The investigators will recruit patients undergoing coronary angiography or coronary computer tomography angiography. Patients' baseline information and facial images will be collected. First, the investigators will explore the facial factors associated with CAD by using artificial intelligence technology to compare facial photographs between patients with CAD and without CAD. Secondary, the investigators will evaluate the dose-response relationship between facial characteristics and CAD. Third, the investigators will establish a CAD risk model based on facial factors, and evaluate the diagnostic effect of the model.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing coronary angiography or coronary computer tomography angiography
* Written informed consent

Exclusion Criteria:

* Prior percutaneous coronary intervention (PCI)
* Prior coronary artery bypass graft (CABG)
* Screening coronary artery disease before treating other heart diseases
* Without blood biochemistry outcome
* With artificially facial alteration (i.e. cosmetic surgery, facial trauma or make-up)
* Other situations which make patients fail to be photographed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who undergo coronary angiography or coronary computer tomography angiography from both resident patients and outpatient.
Sampling Method: Non-Probability Sample
Enrollment: 6864 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity of diagnostic model | at the end of enrollment (6 months)
  The sensitivity of coronary artery diagnostic model assessed in model test group

SECONDARY OUTCOMES:
Specificity of diagnostic model | at the end of enrollment (6 months)
  The specificity of coronary artery diagnostic model assessed in model test group
Specificity of diagnostic model | at the end of enrollment (6 months)
  Area under receiver operating curve (AUC) of diagnostic model assessed in model test group
Positive predictive value (PPV) | at the end of enrollment (6 months)
  PPV of diagnostic model assessed in model test group
Negative predictive value (NPV) | at the end of enrollment (6 months)
  NPV of diagnostic model assessed in model test group
Diagnostic accuracy rate | at the end of enrollment (6 months)
  Diagnostic accuracy rate of diagnostic model assessed in model test group

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Beijing Anzhen hospital, Beijing, Beijing Municipality
  - Fuwai hospital, Beijing, Beijing Municipality
  - Guanganmen Hospital, Chinese Academy of Traditional Chinese Medicine, Beijing, Beijing Municipality
  - Wuhan union hospital, Wuhan, Hubei
  - Xuzhou third people's hospital, Xuzhou, Jiangsu
  - The first affiliated hospital of Dalian medical university, Dalian, Liangning
  - Shanghai East hospital, Shanghai, Shanghai Municipality
  - Shanghai Renji hospital, Shanghai, Shanghai Municipality
  - The fisrt affiliated hospital of Wenzhou medical university, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No